CLINICAL TRIAL: NCT07080047
Title: Mckenzie Technique vs Conventional Therapy in Correcting Lateral Shift in Chronic Lumber Radiculapthy Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01015 Awais Ahmed
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Radiculopathy
Keywords: lumber radiculopathy; radiating pain
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mackenzie exercise for lateral shift (Experimental): Participants in the McKenzie group will perform standing side glide exercises, where they stand perpendicular to a wall (painful side away), press their hips toward the wall, and hold for 2-3 seconds, repeated 30 times. This is followed by five spinal extension repetitions. Sessions will be conducted three times per week for four weeks.
  Interventions: Other: Mackenzie exercise for lateral shift
- Traditional physical therapy (Experimental): Participants in the traditional therapy group will receive posteroanterior lumbar mobilizations (30 repetitions × 3), 10-minute hot pack application, myofascial release of paraspinal muscles, and core stability exercises (plank and bridging). Sessions will be conducted three times per week for four weeks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Mackenzie exercise for lateral shift — Participants in the McKenzie group will perform standing side glide exercises, where they stand perpendicular to a wall (painful side away), press their hips toward the wall, and hold for 2-3 seconds, repeated 30 times
  Arms: Mackenzie exercise for lateral shift
Other: Traditional physical therapy — Participants in the traditional therapy group will receive posteroanterior lumbar mobilizations (30 repetitions × 3), 10-minute hot pack application, myofascial release of paraspinal muscles, and core stability exercises (plank and bridging).
  Arms: Traditional physical therapy

SUMMARY:
Radiculopathy or nerve root pain arises from disc herniation, spinal stenosis/post-operative scarring, radiating down the leg in a dermatomal pattern. Lumbosacral radiculopathy is defined as a "disarticulation of disc components nucleus pulpous or annulus fibrosis beyond the intervertebral disc space. Low back pain (LBP) is one of the most widely recognized conditions that debilitate people's functional capacity in activities of daily living and at work, as well as their general wellbeing and quality of life.

Pain between the buttock and lower edge of the ribs is referred to as low back pain, and it can be classified as acute, sub-acute, or chronic depending on how long it lasts. Acute pain lasts less than four weeks, sub-acute pain lasts more than four but less than twelve weeks and if pain lasts for more than 12 weeks it is chronic LBP. The prevalence of chronic low back pain is steadily rising in today's aging population. Around 80% of the population experience spinal pain sooner or later in life.. The intervertebral disc absorbs physical shock to the backbone; it is composed of two dissimilar tissue layers, an inner layer called the nucleus pulposus and an external layer called the annulus fibrosis. Muscle spasm refers to sustained contraction of a muscle and the increase in chronic tension contributes to pain.

DETAILED DESCRIPTION:
This study is necessary because chronic lumbar radiculopathy often leads to a contralateral lateral shift, causing pain and functional limitations. Traditional physical therapy (TPT) provides general rehabilitation but may not specifically correct this shift. The McKenzie technique (MDT) focuses on self-correction, centralization of symptoms, and postural realignment, making it a potentially superior treatment. However, limited research directly compares McKenzie therapy with TPT for lateral shift correction. This study aims to fill this gap, guiding clinicians toward the most effective rehabilitation approach, improving patient outcomes, and optimizing treatment protocols.• To evaluate the effectiveness of Mackenzie technique versus traditional physical therapy in correcting the lateral shift in patients with chronic lumber radiculopathy.

* To evaluate the effectiveness of Mackenzie technique versus traditional physical therapy in reducing pain in patient with the lateral shift of chronic lumber radiculopathy.
* To determine the effectiveness of Mackenzie technique versus traditional physical therapy in improving range of motion in patients with the lateral shift chronic lumber radiculopathy.
* To determine the effectiveness of Mackenzie technique versus traditional physical therapy in improving functional ability in patients with the lateral shift chronic lumber radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60 years
* Both male and female are included
* Chronic Radiculapathy patients with symptoms lasting from more than 3 months.
* Chronic Radiculapathy patients with contralateral lumber lateral shift.

Exclusion Criteria:

* Fracture, Trauma
* Inflammatory disorder
* Acute disc bulge
* Lumbar instability
* Scoliosis
* Patient with RA and other systemic diseases

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
NPRS | four weeks
  The Numeric Pain Rating Scale (NPRS) is a 0 to 10 self-reported scale used to assess pain intensity, where 0 = no pain and 10 = worst possible pain. It is a simple, reliable tool commonly used in clinical trials to measure pain levels before and after interventions.
Modified Oswestry Disability Index (MODI) | Four weeks
  a validated questionnaire that assesses the degree of disability and functional limitation related to low back pain across daily activities.
Inclinometer | Four weeks
  Lumbar range of motion will be assessed using an inclinometer, a reliable tool that measures spinal movement angles during flexion, extension, and lateral bending.

CONTACTS AND LOCATIONS:
Overall Officials: Zavata Afnan, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Chakdara, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No